CLINICAL TRIAL: NCT04833920
Title: Effect of Motor Cortex Stimulation by Concentric Electrode Transcranial Direct Current Stimulation on Chemotherapy Induced Peripheral Neuropathy
Brief Title: Effect tDCS of Motor Cortex on Chemotherapy Induced Peripheral Neuropathy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Shereen Mamdouh, Associate professor, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 539
Record Dates: First submitted 2021-04-02; First posted 2021-04-06 (Actual); Last update posted 2021-04-06 (Actual); Status verified 2021-04

CONDITIONS: Chemotherapy-induced Peripheral Neuropathy
Keywords: brain stimulation; chemotherapy induced peripheral neuropathy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- active tDCS (Active Comparator): tDCS targeting the primary motor cortex of the contralateral side of the painful side for 20 minute duration for five sessions in five consecutive days
  Interventions: Device: transcranial dirrect current brain stimuation
- sham tDCS (Sham Comparator): tDCS over the primary motor cortex in the same stimulation parameters will be used but the device will be turned off without patient knowledge after 30 seconds
  Interventions: Device: transcranial dirrect current brain stimuation

INTERVENTIONS:
Device: transcranial dirrect current brain stimuation — tDCS (2 mA) targeting the primary motor cortex of the contralateral side of the painful side for 20 minute duration for five sessions in five consecutive days (one session /day),

SUMMARY:
Chemotherapy induced peripheral neuropathy (CIPN) occurs in conjunction with the use of anticancer medication such as vinca alkaloids (including vincristine), taxanes (including paclitaxel), and platinum preparations (including cisplatin and oxaliplatin)

DETAILED DESCRIPTION:
Chemotherapy induced peripheral neuropathy (CIPN) occurs in conjunction with the use of anticancer medication such as vinca alkaloids (including vincristine), taxanes (including paclitaxel), and platinum preparations (including cisplatin and oxaliplatin) . CIPN is one of several long term side effects of anticancer medications that can appear during and after treatment. CIPN symptoms include pain, dysesthesia, motor and sensory disorders. CIPN can also be insufficiently responsive to pharmaceutical therapy similar to other types of refractory neuropathic pain This study is designed to evaluate the effect of two concentric electrode transcranial direct current stimulation (CE-tDCS) over the primary motor cortex (M) in management of chemotherapy induced peripheral neuropathy.

ELIGIBILITY:
Inclusion Criteria:

* any stage of cancer, with a confirmed treatment plan consisting of taxane-based or oxaliplatin-based chemotherapy, neuropathic pain and/or peripheral sensory neuropathy with VAS score ≥ 3 that are resistant to medical treatment

Exclusion Criteria:

* patients with intracranial metallic devices or with pacemakers or any other device. - -W those with extensive myocardial ischemia,
* higher brain dysfunction,
* migraine headache,
* brain cancer or metastasis and
* those known to have epilepsy

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Estimated)
Dates: Start 2021-04-01 (Actual); Primary Completion 2022-01 (Estimated); Study Completion 2022-06 (Estimated)

PRIMARY OUTCOMES:
changes in the visual analogue scale | 0 (prestimulation), on the 5th day, 15th days and one month after the last session
  patient describe his pain scored from 0 to 10 where 0=no pain and 10=the worst pain imaginable

SECONDARY OUTCOMES:
changes in the Leeds Assessment of neuropathic Symptoms and signs (LANSS) | 0 (prestimulation),on the 5th day, 15th days and one month after the last session
  the patients will be asked to describe his pain by answering questions in yes or no; score ≥ 12 suggests neuropathic pain is likely to be involved and score < 12 suggests that neuropathic pain is unlikely to be involved

CONTACTS AND LOCATIONS:
Overall Officials: Shereen M Kamal, Associate Professor, Principal Investigator — Assiut University
Locations (1):
- South Egypt Cancer Institute, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Undecided